CLINICAL TRIAL: NCT04976907
Title: Peri-operative Mobile Application for Contactless Screening and Vital Signs Measurement (MAC-VITAL): A Proof of Concept Trial
Brief Title: Peri-operative Mobile Application for Contactless Screening and Vital Signs Measurement
Acronym: MAC-VITAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nuralogix Corporation (Industry)
Collaborators: University Health Network, Toronto (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Vital Signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perioperative patients: Patients undergoing perioperative assessment of vital signs.
  Interventions: Device: Contactless vital sign information collection

INTERVENTIONS:
Device: Contactless vital sign information collection — Collection of facial blood flow and temperature information via conventional and infrared/thermal video of the face for the purpose of estimating vital signs using machine learning-based computational models.

SUMMARY:
The impact of the coronavirus disease (COVID)-19 pandemic on global healthcare systems has prompted a search for novel tools to stem the tide. New digital health tools can provide possible health solutions in this time of unprecedented medical crisis to mitigate the impact of this pandemic. This proof of concept study will determine the feasibility and effectiveness of implementing a mobile application for contactless screening and vital signs measurement (MAC-VITAL) such as blood pressure (BP), heart rate (HR), respiratory rate (RR), oxyhemoglobin saturation (SpO2), temperature from surgical patients peri-operatively. Contactless measurement of vital signs will bridge the current gap between virtual care and in-person medical assessments.

DETAILED DESCRIPTION:
This study aims to determine whether a mobile app can accurately and reliably measure vital signs without any person to person contact, and the feasibility of implementing it in a peri-operative setting (e.g., during COVID-19). The validity and feasibility of the Anura™ Research app will be assessed during inpatient visits in preparation for and after surgery, and it will be compared with standard medical monitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective surgery under general and/or regional anesthesia
* 18+ years of age

Exclusion Criteria:

* Refusal to consent for the study
* Non-English speaking

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo elective surgery under general and/or regional anesthesia.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure difference from reference measurement (mmHg) | Perioperative
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Diastolic blood pressure difference from reference measurement (mmHg) | Perioperative
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Blood oxygenation (SpO2) difference from reference measurement (% oxyhemoglobin saturation) | Perioperative
  Assessed against standard clinical grade instrument: Finger-based pulse oximeter (% oxyhemoglobin saturation)
Pulse rate difference from reference measurement (beats per minute) | Perioperative
  Assessed against standard clinical grade instrument: Finger-based pulse oximeter (beats per minute)
Teperature difference from reference measurement (degrees Celsius) | Perioperative
  Assessed against standard clinical grade instrument: Forehead digital thermometer (degrees Celsius)
Respiratory rate difference from reference measurement (breaths per minute) | Perioperative
  Assessed against standard clinical grade instrument: Visual count of chest rise and fall (breaths per minute)
Obstacles to using the mobile application | Perioperative
  Characterization of obstacles to the implementation of the mobile app for perioperative vital sign measurements.

SECONDARY OUTCOMES:
Detection rate of clinically meaningful changes of vital signs | Perioperative
  Proportion of clinically meaningful vital sign changes detected postoperatively by the mobile application (relative to vital sign changes detected by standard clinical grade instruments).
Ease of use survey | Perioperative
  Visual analog scale for ease of use.
Satisfaction survey | Perioperative
  Visual analog scale for satisfaction.
Study participation | Perioperative
  Includes: Proportion of patients approached who join the study, proportion of patients who own a mobile phone
Compliance with measurement protocol | Perioperative
  Includes: Proportion of patients who comply with the measurement protocol

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (4):
- Canada (4):
  - Hamilton General Hospital (Hamilton Health Sciences), Hamilton, Ontario
  - Juravinski Hospital (Hamilton Health Sciences), Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario